CLINICAL TRIAL: NCT07048288
Title: Efficacy of Dynamic Exercise and Multi-angle Isometric Exercise Along With Kinesio Taping on Range of Motion, Pain and Functional Disability in Cervical Spondylosis - A Randomized Controlled Trial
Brief Title: Efficacy of Dynamic Exercise and Multi-angle Isometric Exercise in Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AWH/EC/020/2/2023
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Intervention Model Description: A two-arm parallel-group pre-test-post-test design was used in this randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (Experimental): Experimental group 1 received multi-angle isometrics and kinesio taping along with conventional physiotherapy.
  Interventions: Other: Multi-angle isometrics; Other: Kinesio taping; Other: Conventional Physiotherapy
- Experimental Group 2 (Active Comparator): Experimental Group 2 received dynamic exercise and kinesio taping along with conventional physical therapy.
  Interventions: Other: Kinesio taping; Other: Dynamic exercise; Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Multi-angle isometrics — Multi angle exercises include cervical flexion training, Cervical extension training, and Cervical lateral flexion training
  Arms: Experimental Group 1
Other: Kinesio taping — Kinesio taping is a therapeutic technique used in rehabilitation to support muscles and joints without restricting movement.
Other: Dynamic exercise — The dynamic exercise program included dynamic cervical flexion, dynamic cervical extension, and dynamic lateral flexion.
  Arms: Experimental Group 2
Other: Conventional Physiotherapy — Conventional physiotherapy included transcutaneous electrical nerve stimulation

SUMMARY:
Exercises are widely regarded as the primary approach for managing cervical spondylosis. Although several studies have examined the effectiveness of multi-angle isometric exercises and dynamic exercises in patients with cervical spondylosis, their findings have been inconsistent. Further research is warranted to determine whether combining dynamic exercises with Kinesio taping can yield superior therapeutic outcomes. Additionally, there is a lack of comparative studies evaluating the relative benefits of multi-angle isometric versus dynamic exercises for individuals with cervical spondylosis. Therefore, this study aims to compare the efficacy of Multi-angle isometric exercise and Dynamic exercise, along with kinesio taping, in improving range of motion in the cervical spine, reducing pain, and improving functional disability in patients with Cervical Spondylosis. Fifty-two participants were randomly assigned to Experimental Group 1 (EG1) and Experimental Group 2 (EG2), with 26 participants in each group. EG1 received Multi-angle isometrics and Kinesio taping along with conventional physiotherapy, while EG2 received Dynamic exercise and Kinesio taping along with conventional physical therapy. Both groups were treated for 9 weeks. Goniometry and the Neck Pain and disability index were used as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Cervical Spondylosis aged between 30 - 50.
* Both genders.
* Patients with radiological findings of Cervical Spondylosis confirmed by a medical professional.
* Patients without any surgical indication.

Exclusion Criteria:

* Patients with cervical radiculopathy.
* Patients with other cervical spine problems such as; a history of fracture or dislocation, ankylosing spondylitis, congenital cervical anomalies, cervical spine stenosis, cervical spondylotic myelopathy, rheumatoid arthritis, bone tumor, and tuberculosis.
* Patients with pacemakers.
* Patient with psychiatric conditions.
* In cases where the Kinesio taping technique is contraindicated, such as thrombosis, wound, intolerability, allergy to tape, or impaired sensation.
* Patients receiving any form of medications including steroids, NSAIDs or analgesics.
* Patients who do not have good compliance with the intervention or have difficulty in co-operating with the study.
* Patients who cannot read or understand English.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Goniometry | Pre-intervention values were taken before the intervention, and post-intervention values were taken in week 10 (after 9 weeks of treatment).
  Goniometry is the measurement of joint angles using a device called Goniometer. Greater joint angles indicate better treatment outcomes.
Neck Pain and Disability Index | Pre-intervention values were taken before the intervention, and post-intervention values were taken in week 10 (after 9 weeks of treatment).
  The Neck Disability Index (NDI) is a self-report questionnaire designed to measure how neck pain affects a person's ability to manage daily life. Each section has six statements scored from 0 (no disability) to 5 (maximum disability), with a total possible score of 50. The higher the score, the greater the perceived disability.

CONTACTS AND LOCATIONS:
Overall Officials: Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- AWH Special College, Calicut, Kerala, India

IPD SHARING:
Plan to Share IPD: No